CLINICAL TRIAL: NCT07121400
Title: Pedagogical Impact of Different Levels of E-learning Teaching During Anesthesia Residency: a Randomized Clinical Trial
Brief Title: E-learning Teaching During Anesthesia Residency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, jean.selim, Doctor, University Hospital, Rouen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2015-53
Record Dates: First submitted 2025-07-24; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Learning; Anesthesia; Resident Education
Keywords: E-learning; anesthesia residency; resident education; computer-assisted learning; clinical knowledge assessment

STUDY DESIGN:
Intervention Model Description: The participants were randomized into a Passive E-learning group (Pass-EL group) and a Interactive E-learning group (Int-EL group). The Pass-EL group had documents sent by email and the Int-EL group had access to a pedagogical internet platform. A test composed of one clinical case, evaluating the clinical knowledge, and, 15 script concordance tests (SCT), evaluating the clinical reasoning, was conducted before and after e-learning. The outcome of the comparison was the means of the paired within-subject differences (delta) of clinical knowledge scores (pre-and post-test) between the two groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive-E-Learning group (received by email the documents and didn't have access to the platform) (No Intervention): The Passive-E-Learning group only received by email the documents (French experts' recommendations and slide presentation lectures on the management of diabetic patients in anesthesia) and did not have access to the pedagogical internet platform.
- Interactive-E-Learning group (Experimental): The interactive-E-Learning group (Int-EL group) had full access to a pedagogical internet platform with online documents; national experts' recommendations on the management of the diabetic patient in anesthesia, slides presentation lectures on the topic by local university teachers, and, the possibility to contact a virtual mentor (anaesthesiologist of our department) by email for interactive discussion or questions about the topic. The course website was constructed using an online secured program with a unique identification form and password for each resident of the Int-EL group.
  Interventions: Procedure: Interactive e-learning-group

INTERVENTIONS:
Procedure: Interactive e-learning-group — The Interactive-E-learning group had full access to a pedagogical internet platform with online documents; national experts' recommendations on the management of diabetic patients in anesthesia, slide presentation lectures on the topic by local university teachers, and, the possibility to contact a virtual mentor (anaesthesiologist of our department) by email for interactive discussion or questions about the topic.
  Arms: Interactive-E-Learning group

SUMMARY:
E-learning is in expansion although its pedagogical performance has not been validated in the anesthesia residency. E-learning can be divided into passive e-learning; guided e-learning, interactive e-learning, and adaptive e-learning. The objective was to compare the impact of passive e-learning versus interactive e-learning on anesthesia residents' acquisition of theoretical knowledge and clinical reasoning.

DETAILED DESCRIPTION:
The participants first have a pre-test consisting of a clinical case and a script concordance test (SCT). The clinical case was designed to evaluate theoretical clinical knowledge. The clinical case scored 50 points and consisted of 4 open-ended questions (12,5 points for each question) on the management and complications of the diabetic patient in anesthesia. The SCT consisted of 15 questions on the management of the diabetic patient in anesthesia (degenerative neuropathy, ischemic cardiopathy, intubation, management of hyperglycemia, postoperative complications) and was also scored out of 50 points. The participants had 15 minutes for the clinical case and 15 minutes for the SCT.

The pre-test was conducted in a double-blind way, each participant did not know in which group they would be. Each test had a double-blind correction by two senior anesthesiologists. The participants were then randomized to either the Interactive-EL group (Int-EL group) or a Passive-EL group (Pass-EL group).

The Int-EL group had full access to a pedagogical internet platform with online documents; national experts' recommendations on the management of diabetic patients in anesthesia, slide presentation lectures on the topic by local university teachers, and, the possibility to contact a virtual mentor (anaesthesiologist of our department) by email for interactive discussion or questions about the topic.

The Pass-EL group only received by email the documents (French experts' recommendations and slide presentation lectures on the management of diabetic patients in anesthesia) and did not have access to the pedagogical internet platform. The e-learning training period was one month for both groups. The investigators then conducted, in both groups, a post-test composed of the same clinical case and the same SCT.

The time allotted for the post-test was identical to that of the pre-test, and students were not allowed to access external resources during either test.

Each test had a double-blind grading by two senior anesthesiologists.

The tests were developed by two experts in anesthesiology and medical education within our department. The participants in the Pass-EL group had the option to access the platform at the end of the study to complete the e-learning course, should they choose to do so.

ELIGIBILITY:
Inclusion Criteria:

* All anesthesiology residents from first to fourth year in both centers (participants)

Exclusion Criteria:

* Exclusion criteria included residents missing the pre-or post-tests or refusing to participate in the training program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the theoretical clinical knowledge score between the two e-learning groups | One month after pre-test
  The score used was the means of the paired within-subject differences (delta) of clinical knowledge scores (pre-and post-test). The score could range from 0 to 50 points.

SECONDARY OUTCOMES:
The comparison of clinical reasoning scores between the two e-learning groups | one month
  Evaluated by the paired within-subject differences (delta) SCT scores (pre-and post-test). The score could range from 0 to 50 points.
Self-reported difficulty in accessing the pedagogical platform for the Int-EL group and the access to the documents for the Pass-EL group. | one month
  "easy", "medium to difficult" and "difficult"
Self-reported difficulty to validate the MCQs felt by the students of the Int-EL group. | one month
  "easy", "medium to difficult" and "difficult"
Self-reported e-learning usage between the two e-learning groups of the means. | One month
  The reporting time of e-learning usage was in minutes
Student satisfaction score between the two e-learning groups | One month
  Satisfaction score ranging from 0 to 10.

IPD SHARING:
Plan to Share IPD: No